CLINICAL TRIAL: NCT04502680
Title: A Multicenter, Randomized, Open-Label, Phase II Study to Evaluate the Efficacy and Safety of Maintenance Treatment With Eribulin Mesylate Following Standard Adjuvant Chemotherapy in Triple Negative Breast Cancer Patients
Brief Title: Maintenance Treatment With Eribulin Mesylate Versus Observation in Triple Negative Breast Cancer Patients
Acronym: EMBRAVE-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMBRAVE-001
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eribulin Mesylate (Experimental): Patients receive eribulin mesylate following standard adjuvant chemotherapy.
  Interventions: Drug: Eribulin Mesylate
- Observation (No Intervention): Observation. No intervention.

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate 1.4mg/m2, administered intravenously on Days 1 and 8 of each 21 day cycle.
  Other Names: Halaven
  Arms: Eribulin Mesylate

SUMMARY:
This clinical trial is a multicenter, randomized, open-label, phase-II study to evaluate the efficacy and safety of maintenance treatment with eribulin mesylate following standard adjuvant chemotherapy in triple negative breast cancer patients.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) is an aggressive disease with high relapse rates and poor overall survival. This study explores the role of maintenance treatment with eribulin following standard adjuvant chemotherapy in TNBC. Patients will be randomized to receive eribulin mesylate maintenance treatment or observation after standard adjuvant chemotherapy.

The primary objective is to evaluate the disease free survival (DFS). The secondary objective is to evaluate the overall survival (OS), objective response rate (ORR) and the safety of eribulin mesylate maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteers and signs an informed consent form;
* Age ≥18 years old, female;
* The patient was diagnosed as triple-negative breast cancer by histopathology (ER negative (IHC ER positive percentage <1%), PR negative (IHC PR positive percentage <1%), HER2 negative (IHC-/+ or IHC++ but FISH/CISH- )), and there is no evidence of metastasis;
* Patients underwent radical or breast conserving surgery combined with sentinel lymph node biopsy for primary breast cancer. Margins free of disease and ductal carcinoma in-situ (DCIS) are required. Lobular carcinoma is not considered a positive margin.
* For patients who have previously received neoadjuvant therapy for triple-negative breast cancer containing anthracyclines and taxanes, the postoperative efficacy evaluation did not reach pathological complete remission (non-PCR), that is, the primary breast and/or metastatic regional lymph nodes still have histological evidence of malignant tumors other than carcinoma in situ;
* For patients who have not received neoadjuvant therapy for triple-negative breast cancer, ≥1 ipsilateral axillary lymph nodes have pathological tumor involvement after surgery. Or the patient's postoperative lymph nodes are negative, but at least meet one of the following conditions:

  1. Primary invasive tumor size> 2cm in pathology;
  2. Ki-67 index of untreated breast tissue>30%;
  3. The comprehensive score is at least 8 points (Elston and Ellis 1991) according to the improved Bloom-Richardson grading system (also known as the Nottingham scale), which belongs to the 3rd level;
* Physical condition ECOG PS: 0-1;
* Previously received adjuvant chemotherapy consisting of a minimum of 6 courses with anthracyclines combined taxanes;
* Time window between end of adjuvant chemotherapy and study randomization must be less than 8 weeks. In patients receiving adjuvant radiotherapy, time window allowed between last session and randomisation is 4 weeks;
* Laboratory tests meet the following criteria:

  1. Bone marrow function: absolute count of blood neutrophils (ANC) ≥1.5×109/L; platelet (PLT)≥100×109/L; hemoglobin (HB)≥90g/L;
  2. Liver function: serum total bilirubin (STB), combined bilirubin (CB) ≤ upper limit of normal (ULN) *1.5; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN*2.5;
  3. Renal function: serum creatinine (Cr) ≤ ULN; endogenous creatinine clearance (Ccr) ≥ 60 ml / min (calculated using the Cockcroft-Gault formula).

Exclusion Criteria:

* Patients with metastatic breast cancer (including contralateral axillary lymph nodes), inflammatory carcinomas;
* Previous breast cancer history (except for ipsilateral DCIS that only received local treatment ≥5 years ago), malignant tumors of other histological origins (except for non-melanoma skin cancer or cervical carcinoma in situ) unless the patient's tumor had been completely alleviated and had not received treatment for at least 5 years before the enrollment date;
* Major surgery within 4 weeks prior to enrollment, or surgical wounds have not healed;
* Embolization and bleeding occurred within 4 weeks before enrollment;
* Severe cardiovascular disease, including hypertension (BP≥160/95mmHg) uncontrolled by medical treatment, unstable angina, history of myocardial infarction in the past 6 months, congestive heart failure>NYHA II, severe heart rhythm Abnormalities and pericardial effusions;
* Severe infection requires intravenous antibiotic, antifungal or antiviral treatment;
* Suffering from mental illness, poor compliance;
* Researchers believe that it is not suitable for inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 3 years
  DFS was measured from the date of randomization assignment in the intent to treat (ITT) population to loco-regional or distant recurrence, second primary malignancy or death date, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  OS is defined as time to death from any cause.
Objective Response Rate (ORR) | 3 years
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)
The Number of Participants Who Experienced Adverse Events (AE) | 3 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No